CLINICAL TRIAL: NCT03654794
Title: Study of the Cellular Diffusion of Tacrolimus Across the Membrane of Mononuclear Cells
Acronym: DIFF-TAC
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LOC/13-11
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Hemochromatosis
Keywords: Tacrolimus; Pharmacokinetics
MeSH Terms: conditions — Hemochromatosis | interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hemochromatosis: The study is conducted with mononuclear cells obtained from patients undergoing phlebotomy as part of a hemochromatosis treatment.
  The blood samples will be recovered immediately after their completion. 40 mL of blood will be collected and the mononuclear cells separated using a ficoll gradient.
  Cell pharmacokinetics of tacrolimus
  Interventions: Biological: Cell pharmacokinetics of tacrolimus

INTERVENTIONS:
Biological: Cell pharmacokinetics of tacrolimus — Three levels of tacrolimus will be tested. Each aliquot will be supplemented with an amount of tacrolimus to achieve one of these three levels of concentration.
  At 0, 5, 15, 30, 60, 120, 240mn, the samples will be separated into 2 aliquots : one dedicated to the determination of tacrolimus in mononuclear cells, the other dedicated to the determination of calcineurin activity. in mononuclear cells.
  Other Names: Tacrolimus

SUMMARY:
Pharmacokinetics of tacrolimus are highly variable and may result in graft rejection (underdosing) or toxicity (overdosing).

The risk of transplant rejection and the toxicity of tacrolimus can be reduced by pharmacological therapeutic monitoring of the molecule, based on the measurement of residual blood concentrations. Nevertheless, some patients are victims of rejections or toxic signs even though their blood concentrations are in the therapeutic target.

The aim of the study is to describe the pharmacokinetics of tacrolimus diffusion in mononuclear cells as well as the kinetics of effect of the drug on its target protein

DETAILED DESCRIPTION:
Factors responsible for pharmacokinetic variability of tacrolimus are multiple: compliance, diet, drug interactions and also genetic polymorphism of cytochrome P450 3A5 (CYP 3A5) and efflux protein ABCB1 (P-glycoprotein, P-gp).

The mechanism of action of tacrolimus is based on inhibition of calcineurin in T cells. Therefore, tacrolimus intra-lymphocyte concentration may be a finer marker of the risk of transplant rejection or toxicity. The degree of inhibition of calcineurin in the T lymphocyte could also be a pharmacodynamic marker more relevant than the blood concentration. The hypothesis that the ABCB1 efflux pump is the main factor limiting the diffusion of tacrolimus into mononuclear cells is advanced.

The diffusion of tacrolimus into mononuclear cells and the impact of the ABCB1 efflux pump on this diffusion have not been studied to date. The effect kinetics of the drug on calcineurin in mononuclear cells is also unknown.

The aim of the study is to describe the pharmacokinetics of tacrolimus diffusion in mononuclear cells as well as the kinetics of effect of the drug on its target protein: calcineurin in the presence or absence of an efflux pump inhibitor ABCB1 at room temperature and at 4 ° C (in order to inhibit all transport proteins) from blood obtained from 18 patients undergoing bleeding as part of maintenance treatment for hemochromatosis.

ELIGIBILITY:
Inclusion Criteria:

* adult (age > 18 years old);
* phlebotomy as part of the maintenance treatment of hemochromatosis;
* having received the information on the protocol and not having indicated his opposition to participate;
* not receiving immunosuppressive therapy;
* not receiving drug treatment that can induce or inhibit the protein ABCB1 (Rifampicin, Carbamazepine, Phenobarbital, Phenytoin, Efavirenz, Amiodarone, azole antifungals, calcium channel blockers).

Exclusion Criteria:

* participation in another protocol whose procedures are incompatible with the realization of the study;
* adults who are subject to legal protection (protection of justice, guardianship) and persons deprived of their liberty;
* pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing phlebotomy as part of a hemochromatosis treatment
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-10-24 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Diffusion kinetics of tacrolimus in mononuclear cells | At the time of inclusion
  Determination of tacrolimus in mononuclear cells of subjects Tacrolimus will be assayed by mass spectrometry with a limit of quantification of 10 pg / million cells, sufficient to determine the concentrations in the volunteers' blood.

SECONDARY OUTCOMES:
Determination of the activity of calcineurin in mononuclear cells | At the time of inclusion
  These determinations will be carried out by Dr. Benoit Blanchet according to a validated and published method (cf references Blanchet et al, 2003; Blanchet et al, 2006).
  The method is based on high pressure liquid chromatography (HPLC coupled) with spectrophotometric detection.

CONTACTS AND LOCATIONS:
Overall Officials: Florian LEMAITRE, MD, Study Director — Rennes University Hospital
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blanchet B, Hulin A, Duvoux C, Astier A. Determination of serine/threonine protein phosphatase type 2B PP2B in lymphocytes by HPLC. Anal Biochem. 2003 Jan 1;312(1):1-6. doi: 10.1016/s0003-2697(02)00214-2. PMID 12479828
- [Background] Blanchet B, Hulin A, Ghaleh B, Giraudier S, Jouault H, Astier A. Distribution of calcineurin activity in blood cell fractions and impact of tacrolimus inhibition. Fundam Clin Pharmacol. 2006 Apr;20(2):137-44. doi: 10.1111/j.1472-8206.2006.00399.x. PMID 16573714